CLINICAL TRIAL: NCT06336109
Title: The Impacts of Fragmented Sleep on Biomechanics and Pain of the Shoulder and Knee
Brief Title: Fragmented Sleep, Pain, and Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Kristian Kjær Petersen, Associate professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20220063-3
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-04

CONDITIONS: Pain; Healthy; Sleep Disturbance
MeSH Terms: conditions — Pain; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Knee Pain and Shoulder Pain (Experimental): Injection to the infrapatellar fat pad. Will always be administered first.
  Injection to the deltoid muscle. Will always be administered last.
  Interventions: Other: Hypertonic saline knee and shoulder injection

INTERVENTIONS:
Other: Hypertonic saline knee and shoulder injection — 0.25 mL injection with hypertonic saline (7%) in the infrapatellar fat pad.
  1.2 mL injection with hypertonic saline (7%) in the deltoid muscle.

SUMMARY:
This interventional study aims to test the effects of sleep disruption on pain sensitivity and biomechanics in healthy individuals during experimental knee and shoulder pain. The main question the study aims to answer is:

1) Does sleep fragmentation increase experimental knee and shoulder pain and what are the underlying mechanisms?

Participants will receive two injections a) Hypertonic saline (painful) in the knee and b) hypertonic saline (painful) in the upper arm.

DETAILED DESCRIPTION:
This study will include healthy participants for one baseline session and one follow-up session separated by three nights of experimental sleep disruption.

The sleep fragmentation will involve three forced awakenings per night for three consecutive nights between sessions. These awakenings will be planned at 00:00, 02:30, and 05:00.

In each session, the participant will answer questionnaires and have their pain sensitivity assessed using cuff-pressure algometry. Following this, they will first receive a painful saline injection into the infrapatellar fat pad of the knee. After a washout period, they will receive another painful saline injection into the deltoid muscle of the shoulder. For both injections, the pain will be rated on an NRS scale (0 representing 'no pain' and 10 representing 'worst pain imaginable') every 30 seconds, and the distribution will be marked on a body chart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-45 years
* Must have a smartphone available during the experiment

Exclusion Criteria:

* Pregnancy
* Drug addiction, defined as the use of cannabis, opioids, or other drugs
* Previous or current neurologic or musculoskeletal illnesses
* Current pain
* Lack of ability to cooperate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Knee Pain intensity (NRS 0-10) | Baseline (day 1) and follow-up (day 4)
  Pain during intervention is measured continuously every 30 seconds on a numeric rating scale from 0 'no pain' to 10 'the worst pain imaginable'
Shoulder Pain intensity (NRS 0-10) | Baseline (day 1) and follow-up (day 4)
  Pain during intervention is measured continuously every 30 seconds on a numeric rating scale from 0 'no pain' to 10 'the worst pain imaginable'

SECONDARY OUTCOMES:
Pain sensitivity | Baseline (day 1) and follow-up (day 4)
  Cuff-pressure algometry will be used to estimate pressure detection and tolerance thresholds, temporal summation of pain, and conditioned pain modulation.
The Pittsburgh Sleep Quality Index score | Baseline (day 1) and follow-up (day 4)
  19 items summarized to a single score ranging from zero to 21 with higher scores reflecting worse quality of sleep.
The Pain catastrophizing Scale score | Baseline (day 1) and follow-up (day 4)
  13 items summarized to a single score ranging from zero to 52 with higher scores reflecting more catastrophizing.
The Hospital Anxiety and Depression Scale score | Baseline (day 1) and follow-up (day 4)
  14 items summarized into two 7-item subscales measuring symptoms of anxiety and depression. Each subscale score ranges from zero to 21 with higher scores reflecting more severe symptoms.
The Knee injury and Osteoarthritis Outcome Score | Baseline (day 1) and follow-up (day 4)
  42 items divided into five subscales: pain (9 items), activities of daily living (17 items), sport and recreation function (5 items), knee-related quality of life (4 items), and other symptoms (7 items). Each subscale is scored from zero to 100 with higher scores reflecting increased severity of knee problems.
Rapid Assessment of Physical Activity score | Baseline (day 1) and follow-up (day 4)
  9 items scored into summarized categories of either: Sedentary; under-active; under-active regular - light activities; under-active regular; or active.
Pain distribution by number of pixels marked on a body chart | Baseline (day 1) and follow-up (day 4)
  Area marked with pen will be computed into a score of the ratio of pixels marked compared to the total pixels on the body chart.
Video-based motion capture | Baseline (day 1) and follow-up (day 4)
  Video recordings of the participant will be obtained, and will later be processed using machine learning to evaluate the gait pattern.

OTHER OUTCOMES:
Quality of sleep (NRS 0-100) | Baseline (day 1), day 2, day 3 and follow-up (day 4)
  Quality of sleep will be rated from 0 'worst quality imaginable' to 100 'best quality imaginable'.
Level of rest (NRS 0-100) | Baseline (day 1), day 2, day 3 and follow-up (day 4)
  Level of rest will be rated from 0 'not rested at all' to 100 'most rest possible'

CONTACTS AND LOCATIONS:
Overall Officials: Kristian KS Petersen, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No